CLINICAL TRIAL: NCT07032701
Title: Assessing the Impact of a Disposable Negative Pressure Wound Therapy Device on Surgical Wounds of the Lower Extremities Following Mohs Micrographic Surgery
Brief Title: A Disposable Negative Pressure Wound Therapy Device (SNaP) to Promote Wound Healing in the Lower Limbs Following Mohs Micrographic Surgery for Non-melanoma Skin Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-5683; NCI-2025-03606 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-06-16; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Skin Carcinoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods; Aftercare; Negative-Pressure Wound Therapy; Photography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1 (SNaP device dNPWT) (Experimental): Patients undergo dNPWT with SNaP device following SOC Mohs surgery and attend follow-up visits with re-application of SNaP device over 30 minutes QW, as needed until complete wound healing is achieved, for up to 12 weeks. Patients also receive education regarding SNaP device application and informational/educational SNaP device handouts on study.
  Interventions: Other: Educational Intervention; Other: Electronic Health Record Review; Other: Follow-Up Care; Other: Medical Device Usage and Evaluation; Procedure: Negative Pressure Wound Therapy; Other: Photography; Other: Questionnaire Administration
- Group 2 (SOC wound care) (Active Comparator): Patients undergo SOC wound care with non-adherent dressing following SOC Mohs surgery and attend follow-up visits with non-adherent dressing changes over 30 minutes QW, as needed until complete wound healing is achieved, for up to 12 weeks. Patients also receive education on SOC wound dressing changes on study.
  Interventions: Other: Best Practice; Other: Educational Intervention; Other: Electronic Health Record Review; Other: Follow-Up Care; Other: Photography; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Undergo SOC non-adherent dressing wound care
  Other Names: standard of care; standard therapy
  Arms: Group 2 (SOC wound care)
Other: Educational Intervention — Receive SNaP education
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group 1 (SNaP device dNPWT)
Other: Educational Intervention — Receive SOC wound care education
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group 2 (SOC wound care)
Other: Electronic Health Record Review — Ancillary studies
Other: Follow-Up Care — Attend SNaP device follow-up visits
  Arms: Group 1 (SNaP device dNPWT)
Other: Follow-Up Care — Attend SOC wound care follow-up visits
  Arms: Group 2 (SOC wound care)
Other: Medical Device Usage and Evaluation — Undergo dNPWT with SNaP device
  Arms: Group 1 (SNaP device dNPWT)
Procedure: Negative Pressure Wound Therapy — Undergo dNPWT with SNaP device
  Other Names: NPWT; Vacuum-Assisted Wound Closure
  Arms: Group 1 (SNaP device dNPWT)
Other: Photography — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies whether a disposable negative pressure wound therapy (dNPWT) device, SNaP Wound Care System (Ultraportable Mechanically Powered Negative Pressure Wound Therapy) (SNaP), promotes wound healing in the lower limbs in patients that have undergone Mohs micrographic surgery (Mohs surgery) for non-melanoma skin cancer. Mohs surgery is a surgical technique used to treat skin cancer. Individual layers of cancerous tissue are removed and examined under a microscope one at a time until all cancerous tissue has been removed. It is an important part of removing skin cancer, but it often leads to soft-tissue defects and reconstructive challenges, especially in high-tension areas like the lower limbs. Typically, these wounds are managed by leaving them open and allowing them to heal from the base up or are reconstructed by transferring healthy skin from another part of the body. Negative pressure wound therapy (NPWT) is a wound dressing system that continuously or intermittently applies subatmospheric pressure to the surface of a wound to draw out fluid and promote healing. The SNaP device is a dNPWT device for lower leg wound healing designed for increased portability and ease of use outside of a hospital setting. It is a modification of traditional NPWT devices that uses springs to generate pressure, making it lighter and more user-friendly than traditional devices that rely on electrically powered pumps. This may be a more effective way to promote wound healing in the lower limbs following Mohs surgery for non-melanoma skin cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare wound healing duration between the two groups, aiming to provide insights into the potential benefits of dNPWT for lower limb wounds in a clinical setting.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP 1: Patients undergo dNPWT with SNaP device following standard of care (SOC) Mohs surgery and attend follow-up visits with re-application of SNaP device over 30 minutes once a week (QW), as needed until complete wound healing is achieved, for up to 12 weeks. Patients also receive education regarding SNaP device application and informational/educational SNaP device handouts on study.

GROUP 2: Patients undergo SOC wound care with non-adherent dressing following SOC Mohs surgery and attend follow-up visits with non-adherent dressing changes over 30 minutes QW, as needed until complete wound healing is achieved, for up to 12 weeks. Patients also receive education on SOC wound dressing changes on study.

After completion of study intervention, patients are followed up at week 12.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 to 79 years
* Presenting with a lower limb wound following Mohs surgery for non-melanoma skin cancer, designated to heal by secondary intention
* Wound size less than 13 cm x 13 cm
* Patient capable of changing the SNAP-therapy system at home

Exclusion Criteria:

* History of diabetes mellitus
* History of venous insufficiency
* History peripheral arterial disease
* Chronic steroid use (defined as great than 6 weeks) within the last one year
* History of HIV
* History of chemotherapy use within the last one year
* History of smoking exceeding 10 pack-years or current smoker
* History of stroke
* History of deep venous thrombosis
* Active infection
* Allergy to adhesives
* Wounds with visible bone, tendon, ligament, nerve

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2029-01-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Wound healing duration | Up to 12 weeks
  Will be defined as the number of days from surgery to complete wound closure (full re-epithelialization), assessed during follow-up visits. Will be analyzed as a time-to-event variable. To compare the time to wound closure between the SNaP Wound Care System (Ultraportable Mechanically Powered Negative Pressure Wound Therapy) (SNaP) device and standard care groups, Kaplan-Meier survival curves will be generated, which will visually illustrate whether the SNaP device accelerates wound healing. The log-rank test will be used to formally assess whether the difference in healing times between the two groups is statistically significant or if any differences observed could have arisen by random chance. Additionally, a Multivariable Cox proportional hazards model will be employed to adjust for potential confounders (e.g., wound size, patient age, and comorbidities).

SECONDARY OUTCOMES:
Mean time to wound closure | Up to 12 weeks
  Among patients who achieve full healing, the mean time to wound closure will be compared between the SNaP device and standard care groups. If the data are normally distributed, an independent two-sample t-test will be used; otherwise, a Mann-Whitney U test will be applied.
Patient satisfaction | At 12 weeks
  Patient satisfaction will be assessed using standardized questionnaires and analyzed with t-tests or chi-square tests to compare satisfaction levels between the SNaP device and standard care groups. Effect sizes and 95% confidence intervals will be reported to quantify the magnitude of treatment effects for all secondary outcomes.
Wound size progression | Up to 12 weeks
  Wound size progression will be monitored over time and analyzed with repeated measures analysis of variance to assess changes within subjects. Effect sizes and 95% confidence intervals will be reported to quantify the magnitude of treatment effects for all secondary outcomes.
Cosmetic outcomes | At 12 weeks
  Cosmetic outcomes, particularly scar appearance, will be evaluated using the Patient and Observer Scar and Assessment Scale 3.0, with mixed-effects models applied to account for patient variability and treatment effects. Furthermore, a multivariate analysis will be conducted to examine the combined effects of the SNaP device on both wound closure and cosmetic outcomes while adjusting for confounders such as age, comorbidities, and wound size. Effect sizes and 95% confidence intervals will be reported to quantify the magnitude of treatment effects for all secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy C Davis, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States